CLINICAL TRIAL: NCT02346019
Title: Thighplasty of Transfemoral Amputee Residual Limbs to Improve Prosthesis Fit and Patient Functional Outcomes
Brief Title: Thigh Reduction Surgery of Above Knee Amputee Residual Limbs to Improve Prosthesis Fit and Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Todd Kuiken, Director, Center for Bionic Medicine, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00090292
Record Dates: First submitted 2015-01-09; First posted 2015-01-26 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Transfemoral Amputees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical: Medial thighplasty (Experimental): Perform a standard medial thighplasty with our without additional thigh liposuction on up to three obese transfemoral amputee subjects. The surgery will consist of medial excision of excess adipose and cutaneous tissue with circumferential liposuction.
  Interventions: Procedure: Medial thighplasty with or without thigh liposuction

INTERVENTIONS:
Procedure: Medial thighplasty with or without thigh liposuction — Perform a standard medial thighplasty with or without additional thigh liposuction on up to three obese transfemoral amputee subjects. The subjects will be transfemoral amputees who are successful ambulators and have a body mass index (BMI) of 30 or greater with excessive adipose tissue in their residual limb. The surgery will consist of medial excision of excess adipose and cutaneous tissue with circumferential liposuction.

SUMMARY:
The purpose of our study is to improve the fit and function of prosthetic sockets for above the knee amputees through the use of an outpatient thigh reduction surgical procedure.

DETAILED DESCRIPTION:
We will quantify the anatomical distribution of subcutaneous fat, muscle and bone in the residual limb of the transfemoral amputees with an MRI. We will measure the displacement of the socket wall relative to the femur under mechanical loading with x-ray. The functional mobility level of the subject with be quantified via standard clinical and bio mechanical tests. Perform a standard medial thighplasty with our without thigh liposuction. Characterize the post-surgical anatomy, compliance of the residual limb and function of the amputee subjects. After six months, repeat the MRI and xray and compare results. Subject will also complete a questionnaire regarding their views on the outcome of the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Obese transfemoral amputees with a BMI of at least 30.
* Mid to long residual limb, excessive adipose tissue in their residual limb
* Community ambulators
* Adults over the age of 18

Exclusion Criteria:

* Amputation due to vascular disease or diabetes
* Cognitive impairments that would interfere with the protocol or patient safety
* Systemic disease that is not stable or would significantly increase the risk of complications with surgery
* Chronic wounds
* People who do not ambulate on a daily basis
* Children under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-08; Primary Completion 2019-08 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Assess compliance of residual limb in the socket, which will improve the fit and comfort of the prosthesis. | Pre surgery and 6 months post surgery
  We will measure the compliance of their residual limb by the displacement of the socket wall relative to the femur under mechanical loading with X-ray. The subjects will adjust their foot placement, limb loading and muscle contractions to achieve up to 8 specified force/torque levels (as measured by a 6 degree-of-freedom load cell located in series with their pylon and socket), which correspond to forces and torques that are typical of over ground walking and standing postures and are scaled for their body weight. For each force/torque level, static X-ray scans of locations of the prosthetic socket wall and residual limb femur will be acquired.

SECONDARY OUTCOMES:
Assess walking endurance | Pre surgery and 6 months post surgery
  Complete 6 minute walk test over level ground as metabolic energy consumption and heart rate our monitored. Subjects may wear a portable, commercially available metabolic measurement system so that their metabolic energy expenditure may be calculated after the experiment.
Assess balance stability | Pre surgery and 6 months post surgery
  Complete the 4 square step test as a clinical test of the ability to change directions while stepping.

CONTACTS AND LOCATIONS:
Overall Officials: Todd A Kuiken, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States